CLINICAL TRIAL: NCT02773186
Title: Cerebral Oximetry With Near-infrared Spectroscopy and Negative Postoperative Behavioral Changes in Pediatric Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Estefanía Gomez Pesquera, MD Anesthesiologist, Hospital Clínico Universitario de Valladolid
Other Study IDs: NPOBC
Record Dates: First submitted 2016-04-21; First posted 2016-05-16 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Cognitive Dysfunction
Keywords: postoperative; behavioral changes
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: monitoring cerebral oxygen saturation — Children undergoing urological surgery also required of locoregional blockade. Anesthetic induction was achieved with high concentration sevoflurane 6-8% (Sevorane®, Abbvie) and oxygen 50%. Anesthetic maintenance was done with sevoflurane 2-3%, 50% O2/air mixture, fentanyl 1 µg.kg.-1 iv, and rocuronium 0.3 µg.kg.-1 iv if required. Electrocardiogram (ECG), non-invasive arterial pressure, pulse oximetry, end-tidal carbon dioxide and cerebral NIRS oximetry was monitoring by using an INVOSTM5100 (Somanetics Corporation, Troy, MI, USA).

SUMMARY:
The main objective of the present study was to evaluate whether cerebral oxygen saturation is associated with an increase of NPOBC in pediatric patients undergoing major surgery.

DETAILED DESCRIPTION:
This prospective and observational study involved consecutive patients aged between 2 and 12 years undergoing a major surgery using general anesthesia. Cerebral oxygen saturation, non-invasive arterial pressure, pulse oximetry, and heart rate were recorded at the following stages of the surgical intervention: baseline, induction, intubation, surgical incision, end of surgery, and extubation. Preoperative anxiety was evaluated by using the modified Yale Preoperative Anxiety Scale, and NPOBC was determined by using the Post-Hospital Behaviour Questionnaire on 7th and 28th postoperative days. A logistic regression was created to identify factors associated with the development of NPOBC

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 2 and 12 years undergoing major surgery using general anesthesia.

Exclusion Criteria:

* Children aged below 2 or over 12.
* Neuropsychiatric disorder, or undergoing an emergency surgery.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This prospective and observational study involved consecutive patients aged between 2 and 12 years undergoing a major surgery using general anesthesia.Children undergoing urological and general surgery also required of locoregional blockade. Anesthetic induction was achieved with high concentration sevoflurane 6-8% (Sevorane®, Abbvie) and oxygen 50%. Anesthetic maintenance was done with sevoflurane 2-3%, 50% O2/air mixture, fentanyl 1 µg.kg.-1 iv, and rocuronium 0.3 µg.kg.-1 iv if required. Electrocardiogram (ECG), non-invasive arterial pressure, pulse oximetry, end-tidal carbon dioxide and cerebral NIRS oximetry was monitoring by using an INVOSTM5100 (Somanetics Corporation, Troy, MI, USA)
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Negative Postoperative Behavioral Changes | on 7th and 28th postoperative days
  NPOBC was measured by using thePost-Hospital Behaviour Questionnaire.

SECONDARY OUTCOMES:
Number of children with cerebral desaturation and NPOBC | on 7th and 28th postoperative days
  Cerebral oxygen saturation was monitoring by using the monitor INVOS 5100

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tamayo Gómez, MD PhD, Study Director

IPD SHARING:
Plan to Share IPD: Undecided
there is not plan by the moment